CLINICAL TRIAL: NCT06137339
Title: AvoCog - The Effect of Daily Avocado Intake on Cognitive Function in Older Adults
Acronym: AvoCog
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Collaborators: Avocado Nutrition Center (Unknown)
Responsible Party: Principal Investigator, Matthew Taylor, Dr. Matthew K Taylor, PhD, RD, University of Kansas Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 00150975
Record Dates: First submitted 2023-11-13; First posted 2023-11-18 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Brain Aging
Keywords: Older Adults; Brain Health; Avocado; Brain Imaging; Cognition; Dietary Intervention

STUDY DESIGN:
Intervention Model Description: Study participants will be randomly assigned equally to either the intervention or the control group.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Participants cannot be blinded to their allocation in order to follow the study protocol. Investigator and Outcomes Assessor will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Avocado Group (Experimental): Participants will consume 1 avocado per day and receive education to maintain usual caloric intake for 12 weeks and participate in 4 study visits.
  Interventions: Other: Avocado Group
- No Diet Modification Group (No Intervention): Participants will continue their normal dietary pattern for 12 weeks and participate in 4 study visits.

INTERVENTIONS:
Other: Avocado Group — Participants will consume provided avocados daily and track consumption for the duration of the study. Participants will be adding avocados to their diet and will receive education on maintaining usual diet.
  Arms: Avocado Group

SUMMARY:
The goal of this clinical trial is to determine if adding avocados to the diet of impacts cognition in 70 older adults, age 65-85, without dementia. We will test for change in functional MRI, cognitive performance, and brain blood flow. Intervention group participants will be asked to consume 1 avocado per day for 12 weeks. Participants in the control group will be asked to continue their normal intake for 12 weeks. Throughout the study, participants will be asked to perform cognitive tests, MRI, blood tests, and questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged 65-85 years
* Good general health with no concomitant disease
* BMI 18.5 - 35 kg/m2
* Mini Mental State Exam ≥26
* Reports consuming ≤2 medium avocados per month
* Reports consuming ≤3 servings of carotenoid-rich foods per week and ≤3 servings of fruits and vegetables per day
* Skin carotenoid content <400

Exclusion Criteria:

* Unwilling or unable to consume avocado
* Latex allergy
* Consistently taking lutein + zeaxanthin supplements
* Skin carotenoid content ≥400
* Central neurological disease such as Alzheimer's disease, Parkinson's disease, multiple sclerosis, stroke, brain tumor, etc.
* Serious medical risk: cancer requiring chemotherapy or radiation within the past 5 years, recent cardiac event (i.e. heart attack, etc.)
* Diabetes mellitus or uncontrolled hypertension
* Use of psychoactive or investigational medications
* Consumption of ≥3 alcoholic drinks per day or substance abuse
* Unable to undergo MRI

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-04-09 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change in brain activity | Baseline and 12 weeks
  MRI will be used to measure changes in brain activity during resting state, a working memory task, and executive function task.

SECONDARY OUTCOMES:
Changes in cerebral blood flow | Baseline and 12 weeks
  MRI will be used to measure change in cerebral blood flow.
Changes in memory and executive function | Baseline and 12 weeks
  NIH Toolbox will be used to measure change in cognition throughout the study.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: No